CLINICAL TRIAL: NCT01597908
Title: A Phase III, Randomised, Open-label Study Comparing the Combination of the BRAF Inhibitor, Dabrafenib and the MEK Inhibitor, Trametinib to the BRAF Inhibitor Vemurafenib in Subjects With Unresectable (Stage IIIc) or Metastatic (Stage IV) BRAF V600E/K Mutation Positive Cutaneous Melanoma
Brief Title: Dabrafenib Plus Trametinib vs Vemurafenib Alone in Unresectable or Metastatic BRAF V600E/K Cutaneous Melanoma
Acronym: COMBI-v
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116513; CDRB436B2302 (Other: Novartis); 2011-006088-23 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
Keywords: BRAF inhibitor; Metastatic Melanoma; Cancer; MEK inhibitor
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — dabrafenib; Vemurafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabrafenib plus Trametinib (Experimental): BRAF inhibitor plus MEK inhibitor
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Vemurafenib (Active Comparator): BRAF inhibitor
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib 150 mg twice daily orally
  Other Names: GSK2118436
  Arms: Dabrafenib plus Trametinib
Drug: Vemurafenib — Vemurafenib 960 mg twice daily orally
  Other Names: Monotherapy
  Arms: Vemurafenib
Drug: Trametinib — Trametinib 2 mg once daily orally
  Other Names: GSK1120212
  Arms: Dabrafenib plus Trametinib

SUMMARY:
This was a two-arm, open-label, randomized, Phase III study comparing dabrafenib (GSK2118436) and trametinib (GSK1120212) combination therapy with vemurafenib.

DETAILED DESCRIPTION:
Screening/Subject eligibility: Subjects with histologically confirmed cutaneous melanoma that was either unresectable or metastatic (Stages IIIC or IV), were screened for eligibility. Eligible subjects were BRAF V600E or V600K mutation positive. Subjects who had prior systemic anti-cancer treatment in the advanced or metastatic setting were not eligible although prior systemic treatment in the adjuvant setting was allowed.

Randomization: A total of 704 subjects were randomized in a ratio of 1:1 to receive combination therapy (352 subjects) or vemurafenib treatment (352 subjects). Subjects were stratified by LDH level (> the ULN versus =< ULN) and BRAF mutation (V600E versus V600K).

Study treatment: Dabrafenib and trametinib were administered orally at their recommended doses of 150 mg b.i.d. and 2.0 mg once daily, respectively. Subjects randomized in the combination therapy arm received both the agents. Subjects randomized in the vemurafenib arm received vemurafenib at the recommended dose of 960 mg orally b.i.d. Subjects in both the arms continued treatment until disease progression, death, unacceptable toxicity, or withdrawal of consent. The protocol was amended on 07-Aug-2014 which allowed subjects who were still receiving vemurafenib to cross over to the dabrafenib and trametinib combination arm, including those subjects who were still receiving vemurafenib monotherapy treatment after disease progression. A washout period of a minimum of 7 days was considered prior to initiating dabrafenib in combination with trametinib. Subjects who experienced disease progression on the vemurafenib monotherapy arm, discontinued vemurafenib monotherapy, and subsequently received another anticancer therapy were ineligible for cross over to the dabrafenib and trametinib combination arm.

Follow-up/Study closure: After study treatment discontinuation, subjects were followed for survival and disease progression as applicable. This study completed once all the subjects had at least the 5-years of follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* >= 18 years of age
* Stage IIIc or Stage IV BRAF V600E/K cutaneous melanoma
* Measurable disease according to RECIST 1.1
* Women of childbearing potential with negative serum pregnancy test prior to randomisation
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Adequate baseline organ function

Key Exclusion Criteria:

* Any prior use of a BRAF or MEK inhibitor
* Prior systemic anti-cancer treatment in the advanced or metastatic setting; prior systemic treatment in the adjuvant setting is allowed
* History of another malignancy (except subjects who have been disease free for 3 years or with a history of completely resected non-melanoma skin cancer)
* Known HIV, HBV, HCV infection (except chronic or cleared HBV and HCV infection which will be allowed)
* Brain metastases (except if all known lesions were previously treated with surgery or stereotactic radiosurgery and lesions, if still present, are confirmed stable for >= 12 weeks prior to randomisation or if no longer present are confirmed no evidence of disease for >= 12 weeks, and are asymptomatic with no corticosteroid requirements for >= 4 weeks prior to randomisation, and no enzyme inducing anticonvulsants for >= 4 weeks prior to randomisation
* History or evidence of cardiovascular risk (LVEF < LLN; QTcB >= 480 msec; blood pressure or systolic >=140 mmHg or diastolic >= 90 mmHg which cannot be controlled by anti-hypertensive therapy)
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2014-04-17 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (186):
- United States (33):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Vallejo, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami Beach, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Bend, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Viedma, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
- Australia (9):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (4):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (7):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Wilrijk
- Brazil (3):
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, Sao Paulo - SP
- Canada (11):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Kingston, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (4):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Zlín
- Denmark (3):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense
- Finland (4):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (11):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Villejuif
- Germany (23):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Heilbronn, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Buxtehude, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Gera, Thuringia
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Szeged
- Ireland (3):
  - Novartis Investigative Site, Co.Cork
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (7):
  - Novartis Investigative Site, Napoli, Campania
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Pisa, Tuscany
  - Novartis Investigative Site, Padua, Veneto
- Netherlands (5):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Rotterdam
- New Zealand (2):
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Newtown, Wellington
- Norway (3):
  - Novartis Investigative Site, Kristiansand
  - Novartis Investigative Site, Lorenskog
  - Novartis Investigative Site, Oslo
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Russia (6):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Magnitogorsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
- South Korea (2):
  - Novartis Investigative Site, Goyang-si, Gyeonggi-Do
  - Novartis Investigative Site, Seoul
- Spain (7):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Valencia
- Sweden (2):
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Umeå
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Ukraine (7):
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Sumy
  - Novartis Investigative Site, Uzhhorod
- United Kingdom (6):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Schadendorf D, Robert C, Dummer R, Flaherty KT, Tawbi HA, Menzies AM, Banerjee H, Lau M, Long GV. Pyrexia in patients treated with dabrafenib plus trametinib across clinical trials in BRAF-mutant cancers. Eur J Cancer. 2021 Aug;153:234-241. doi: 10.1016/j.ejca.2021.05.005. Epub 2021 Jul 2. PMID 34225229
- [Derived] Robert C, Grob JJ, Stroyakovskiy D, Karaszewska B, Hauschild A, Levchenko E, Chiarion Sileni V, Schachter J, Garbe C, Bondarenko I, Gogas H, Mandala M, Haanen JBAG, Lebbe C, Mackiewicz A, Rutkowski P, Nathan PD, Ribas A, Davies MA, Flaherty KT, Burgess P, Tan M, Gasal E, Voi M, Schadendorf D, Long GV. Five-Year Outcomes with Dabrafenib plus Trametinib in Metastatic Melanoma. N Engl J Med. 2019 Aug 15;381(7):626-636. doi: 10.1056/NEJMoa1904059. Epub 2019 Jun 4. PMID 31166680
- [Derived] Long GV, Grob JJ, Nathan P, Ribas A, Robert C, Schadendorf D, Lane SR, Mak C, Legenne P, Flaherty KT, Davies MA. Factors predictive of response, disease progression, and overall survival after dabrafenib and trametinib combination treatment: a pooled analysis of individual patient data from randomised trials. Lancet Oncol. 2016 Dec;17(12):1743-1754. doi: 10.1016/S1470-2045(16)30578-2. Epub 2016 Nov 16. PMID 27864013
- [Derived] Grob JJ, Amonkar MM, Karaszewska B, Schachter J, Dummer R, Mackiewicz A, Stroyakovskiy D, Drucis K, Grange F, Chiarion-Sileni V, Rutkowski P, Lichinitser M, Levchenko E, Wolter P, Hauschild A, Long GV, Nathan P, Ribas A, Flaherty K, Sun P, Legos JJ, McDowell DO, Mookerjee B, Schadendorf D, Robert C. Comparison of dabrafenib and trametinib combination therapy with vemurafenib monotherapy on health-related quality of life in patients with unresectable or metastatic cutaneous BRAF Val600-mutation-positive melanoma (COMBI-v): results of a phase 3, open-label, randomised trial. Lancet Oncol. 2015 Oct;16(13):1389-98. doi: 10.1016/S1470-2045(15)00087-X. PMID 26433819
- [Derived] Robert C, Karaszewska B, Schachter J, Rutkowski P, Mackiewicz A, Stroiakovski D, Lichinitser M, Dummer R, Grange F, Mortier L, Chiarion-Sileni V, Drucis K, Krajsova I, Hauschild A, Lorigan P, Wolter P, Long GV, Flaherty K, Nathan P, Ribas A, Martin AM, Sun P, Crist W, Legos J, Rubin SD, Little SM, Schadendorf D. Improved overall survival in melanoma with combined dabrafenib and trametinib. N Engl J Med. 2015 Jan 1;372(1):30-9. doi: 10.1056/NEJMoa1412690. Epub 2014 Nov 16. PMID 25399551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 207 centers in 28 countries worldwide (Argentina, Australia, Austria, Belgium, Brazil, Canada, Czech Republic, Denmark, Finland, France, Germany, Hungary, Ireland, Israel, Italy, South Korea, Netherlands, New Zealand, Norway, Poland, Russian Federation, Spain, Sweden,Switzerland, Taiwan, Ukraine, UK and USA).
Pre-assignment Details: 694 subjects were planned and 704 subjects (352 each in combination therapy arm and vemurafenib monotherapy arm) were actually randomized and analyzed. Subjects were stratified by LDH level (> the ULN versus ≤ ULN) and BRAF mutation (V600E versus V600K).
Groups:
- Dabrafenib Plus Trametinib: Dabrafenib 150 milligrams (mg) orally twice daily (BID) and Trametinib 2 mg orally once daily until disease progression, death, unacceptable toxicity, or withdrawal of consent.
- Vemurafenib: Vemurafenib 960 mg orally BID until disease progression, death, unacceptable toxicity, or withdrawal of consent.
- Crossover Dabrafenib Plus Trametinib: With Protocol Amendment 7, patients still receiving study treatment on the Vemurafenib monotherapy arm were allowed to cross over to the Dabrafenib and Trametinib combination arm.
Period: Randomized Phase
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib | Crossover Dabrafenib Plus Trametinib
Started (All randomized patients included into Intent-to-Treat (ITT) population.) | 352 | 352 | 0
Safety Set (All patients who received at least one dose of study treatment) | 350 | 349 | 0
Completed (ongoing status (incomplete end-of-study data and never received study treatment)) | 1 | 0 | 0
Not Completed | 351 | 352 | 0
Not completed — Death | 217 | 238 | 0
Not completed — Sponsor Decision | 93 | 39 | 0
Not completed — Lost to Follow-up | 9 | 16 | 0
Not completed — Physician Decision | 6 | 3 | 0
Not completed — Withdrawal by Subject | 26 | 22 | 0
Not completed — Crossover to Dabrafenib&Trametinib | 0 | 34 | 0
Period: Crossover Phase
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib | Crossover Dabrafenib Plus Trametinib
Started (All crossover randomized patients included into ITT & Safety Sets) | 0 | 0 | 34
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 34
Not completed — Death | 0 | 0 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Sponsor Decision | 0 | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib | Total
Number analyzed (Participants) | 352 | 352 | 704
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (13.83) | 54.3 (14.06) | 54.2 (13.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 172 | 316
  Male | 208 | 180 | 388
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 8 | 8 | 16
  White - Arabic/North African Heritage | 4 | 2 | 6
  White - White/Caucasian/European Heritage | 339 | 339 | 678
  White - Mixed Race | 1 | 0 | 1
  Mixed Race | 0 | 1 | 1
  African American/African Heritage | 0 | 1 | 1
  American Indian or Alaskan Native | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the interval of time between the date of randomization and the date of death due to any cause. For patients who did not die, OS was censored at the date of last contact.
Time Frame: From the date of randomization until date of death due to any cause (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib
Number analyzed (Participants) | 352 | 352
Months | 26.0 [22.1 to 33.8] | 17.8 [15.6 to 20.7]
Statistical Analysis 1: Comparison: Dabrafenib Plus Trametinib vs Vemurafenib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.58 to 0.83] — Hazard ratios are estimated using a Pike estimator

2. Secondary Outcome: Progression-Free Survival (PFS), as Assessed by the Investigator
Description: Progression-free survival (PFS) was defined as the interval of time between the date of randomization and the first documented occurrence of disease progression or death due to any cause. PFS for investigator-assessed response was summarized per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1, which is a set of published rules defining when cancer patients improve (respond), stay the same (stabilize), or worsen (progress) during treatment. Disease progression was defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 millimeters (mm) or the appearance of at least 1 new lesion, or the worsening of non-target lesions significant enough to require study treatment discontinuation.
Time Frame: From randomization until the earliest date of disease progression (PD) or death due to any cause (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib
Number analyzed (Participants) | 352 | 352
Months | 12.1 [9.7 to 14.7] | 7.3 [6.0 to 8.1]
Statistical Analysis 1: Comparison: Dabrafenib Plus Trametinib vs Vemurafenib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.52 to 0.73] — Hazard ratios are estimated using a Pike estimator

3. Secondary Outcome: Overall Response Rate (ORR) During Randomized Phase, as Assessed by the Investigator
Description: Overall response was defined as the percentage of confirmed responders (complete response [CR] + partial response [PR] per RECIST, Version 1.1) as summarized by Investigator assessment. CR was defined as the disappearance of all evidence of target lesions. PR was defined as at least a 30% reduction from Baseline in the sum of the longest diameter (LD) of all target lesions. Data were reported as those participants with measureable disease at Baseline.
Time Frame: From randomization until the first documented complete response or partial response (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population. Only participants with measurable disease at baseline were included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib
Number analyzed (Participants) | 351 | 350
Percentage of Participants | 68 [62.3 to 72.4] | 53 [47.2 to 57.9]

4. Secondary Outcome: Duration of Response (DOR), as Assessed by the Investigator
Description: Duration of Response (DOR) was defined as the time from the first documented evidence of a CR (disappearance of all evidence of target lesions) or a PR (at least a 30% reduction from Baseline in the sum of the longest diameter of all target lesions) until disease progression or death due to any cause. PD was defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5 mm or the appearance of at least1 new lesion, or the worsening of non-target lesions significant enough to require study treatment discontinuation. Data were summarized per RECIST, Version 1.1.
Time Frame: From the time of the first documented response (CR or PR) until disease progression (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population. Only participants with confirmed response by RECIST version 1.1 were included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib
Number analyzed (Participants) | 237 | 185
Months | 13.8 [11.3 to 18.6] | 8.5 [7.4 to 9.3]
Statistical Analysis 1: Comparison: Dabrafenib Plus Trametinib vs Vemurafenib; Test type: Superiority or Other; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.51 to 0.81]

5. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from screening visit up to the first day of treatment, for a maximum duration of 28 days. Patients who died during the screening period are considered as screen failure.
  On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 81.1 months (treatment duration ranged from 0.1 to 80.1 months).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 6 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 28 days before Day 1 (Screening), up to 81.1 months (on-treatment), up to approximately 6 years (study duration)
Population: Clinical database population; all treated patients and patients who died during screening.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Dabrafenib + Trametinib: With Protocol Amendment 7, patients still receiving study treatment on the Vemurafenib monotherapy arm were allowed to cross over to the Dabrafenib and Trametinib combination arm.
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib | Crossover Dabrafenib + Trametinib
Number analyzed (Participants) | 351 | 349 | 34
Participants
  Pre-treatment deaths | 1 | 0 | 0
  On-treatment deaths | 44 | 47 | 2
  Post-treatment deaths | 172 | 191 | 9
  All deaths | 216 | 238 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of 81.1 months (treatment duration ranged from 0.1 to 80.1 months). In addition, new malignancies and AEs possibly related to study treatment were collected up to approximately 6 years
Description: Any clinically significant sign or symptom that occurs during the study treatment and 30 days post treatment follow up. In addition, new malignancies and AEs possibly related to study treatment were collected even if they occurred more than 30 days post-treatment.
Groups:
- All Patients: All randomized patients who received at least one dose of study treatment.
Arm/Group | Dabrafenib Plus Trametinib | Vemurafenib | Crossover Dabrafenib Plus Trametinib | All Patients
All-Cause Mortality (participants affected / at risk) | 216/350 | 238/349 | 11/34 | 465/699
Serious Adverse Events (participants affected / at risk) | 172/350 | 139/349 | 15/34 | 319/699
Other Adverse Events (participants affected / at risk) | 338/350 | 341/349 | 32/34 | 679/699
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib Plus Trametinib (N=350) | Vemurafenib (N=349) | Crossover Dabrafenib Plus Trametinib (N=34) | All Patients (N=699)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 1 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 4 | 0 | 7
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2 | 0 | 4
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 5 | 0 | 5
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 2
Cataract (Eye disorders) | 1 | 0 | 0 | 1
Chorioretinopathy (Eye disorders) | 2 | 1 | 0 | 3
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0 | 1
Retinal degeneration (Eye disorders) | 0 | 1 | 0 | 1
Retinal tear (Eye disorders) | 1 | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 2 | 0 | 2
Uveitis (Eye disorders) | 1 | 1 | 0 | 2
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 6
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 8 | 1 | 0 | 9
Asthenia (General disorders) | 3 | 0 | 0 | 3
Chest pain (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 14 | 0 | 0 | 14
Fatigue (General disorders) | 2 | 1 | 1 | 4
General physical health deterioration (General disorders) | 0 | 1 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 3 | 0 | 0 | 3
Malaise (General disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 55 | 6 | 0 | 61
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 2 | 0 | 6
Cholelithiasis (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Abscess soft tissue (Infections and infestations) | 1 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 5 | 1 | 0 | 6
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 1
Corneal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0 | 2
Erysipelas (Infections and infestations) | 4 | 0 | 0 | 4
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Gastrointestinal infection (Infections and infestations) | 3 | 2 | 0 | 5
Haematoma infection (Infections and infestations) | 1 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 1
Infection (Infections and infestations) | 2 | 1 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Meningitis (Infections and infestations) | 0 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 6 | 1 | 10
Post procedural infection (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 3 | 0 | 1 | 4
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 10 | 1 | 1 | 12
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 9 | 0 | 15
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 0 | 8
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 6 | 0 | 8
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 0 | 3
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 3
Ejection fraction decreased (Investigations) | 31 | 1 | 2 | 34
Hepatic enzyme increased (Investigations) | 4 | 6 | 0 | 10
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 1
Troponin I increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 2 | 0 | 10
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 5 | 2 | 20
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0 | 5
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 23 | 1 | 26
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7 | 0 | 9
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 27 | 0 | 30
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 30 | 0 | 33
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 3 | 1 | 0 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 1 | 1 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 0 | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 2 | 1 | 0 | 3
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 3
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 0 | 0 | 4
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 2
Hypotension (Vascular disorders) | 5 | 0 | 0 | 5
Lymphocele (Vascular disorders) | 0 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 1
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib Plus Trametinib (N=350) | Vemurafenib (N=349) | Crossover Dabrafenib Plus Trametinib (N=34) | All Patients (N=699)
Anaemia (Blood and lymphatic system disorders) | 29 | 20 | 3 | 52
Leukopenia (Blood and lymphatic system disorders) | 17 | 7 | 6 | 29
Lymphopenia (Blood and lymphatic system disorders) | 9 | 9 | 2 | 20
Neutropenia (Blood and lymphatic system disorders) | 37 | 6 | 9 | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 2 | 3 | 16
Tinnitus (Ear and labyrinth disorders) | 5 | 3 | 2 | 10
Vision blurred (Eye disorders) | 23 | 18 | 1 | 42
Abdominal pain (Gastrointestinal disorders) | 41 | 33 | 3 | 75
Abdominal pain upper (Gastrointestinal disorders) | 38 | 36 | 4 | 78
Constipation (Gastrointestinal disorders) | 58 | 25 | 7 | 89
Diarrhoea (Gastrointestinal disorders) | 131 | 137 | 5 | 268
Dry mouth (Gastrointestinal disorders) | 27 | 8 | 1 | 36
Dyspepsia (Gastrointestinal disorders) | 20 | 15 | 3 | 37
Haemorrhoids (Gastrointestinal disorders) | 4 | 7 | 3 | 14
Nausea (Gastrointestinal disorders) | 125 | 131 | 8 | 261
Vomiting (Gastrointestinal disorders) | 111 | 57 | 4 | 172
Asthenia (General disorders) | 65 | 62 | 8 | 131
Chills (General disorders) | 113 | 28 | 6 | 147
Fatigue (General disorders) | 116 | 116 | 1 | 232
Hypothermia (General disorders) | 2 | 1 | 2 | 4
Influenza like illness (General disorders) | 36 | 13 | 2 | 51
Malaise (General disorders) | 16 | 8 | 2 | 24
Oedema peripheral (General disorders) | 61 | 45 | 3 | 108
Pain (General disorders) | 18 | 15 | 2 | 35
Peripheral swelling (General disorders) | 25 | 12 | 3 | 40
Pyrexia (General disorders) | 184 | 72 | 16 | 267
Angular cheilitis (Infections and infestations) | 3 | 0 | 2 | 5
Conjunctivitis (Infections and infestations) | 14 | 37 | 1 | 52
Folliculitis (Infections and infestations) | 18 | 25 | 1 | 43
Influenza (Infections and infestations) | 31 | 9 | 2 | 41
Nasopharyngitis (Infections and infestations) | 64 | 32 | 6 | 100
Onychomycosis (Infections and infestations) | 4 | 1 | 2 | 7
Pharyngitis (Infections and infestations) | 19 | 7 | 1 | 27
Pneumonia (Infections and infestations) | 4 | 1 | 4 | 9
Rhinitis (Infections and infestations) | 14 | 8 | 2 | 24
Upper respiratory tract infection (Infections and infestations) | 23 | 14 | 3 | 40
Urinary tract infection (Infections and infestations) | 31 | 7 | 3 | 41
Fall (Injury, poisoning and procedural complications) | 6 | 5 | 2 | 12
Sunburn (Injury, poisoning and procedural complications) | 5 | 47 | 0 | 52
Alanine aminotransferase increased (Investigations) | 54 | 54 | 2 | 110
Aspartate aminotransferase increased (Investigations) | 47 | 42 | 3 | 92
Blood alkaline phosphatase increased (Investigations) | 30 | 29 | 0 | 59
Blood creatine phosphokinase increased (Investigations) | 12 | 4 | 5 | 20
Blood creatinine increased (Investigations) | 16 | 36 | 2 | 53
Blood lactate dehydrogenase increased (Investigations) | 23 | 9 | 1 | 33
C-reactive protein increased (Investigations) | 12 | 1 | 2 | 15
Gamma-glutamyltransferase increased (Investigations) | 45 | 35 | 1 | 81
Neutrophil count decreased (Investigations) | 15 | 1 | 2 | 18
Weight decreased (Investigations) | 21 | 42 | 1 | 64
White blood cell count decreased (Investigations) | 13 | 3 | 2 | 18
Decreased appetite (Metabolism and nutrition disorders) | 47 | 72 | 6 | 123
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 12 | 3 | 35
Increased appetite (Metabolism and nutrition disorders) | 2 | 1 | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 104 | 182 | 9 | 288
Back pain (Musculoskeletal and connective tissue disorders) | 43 | 29 | 5 | 77
Muscle spasms (Musculoskeletal and connective tissue disorders) | 47 | 13 | 4 | 63
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 | 10 | 0 | 29
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 27 | 4 | 54
Myalgia (Musculoskeletal and connective tissue disorders) | 76 | 56 | 8 | 134
Pain in extremity (Musculoskeletal and connective tissue disorders) | 50 | 42 | 2 | 94
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 21 | 0 | 23
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 85 | 1 | 95
Balance disorder (Nervous system disorders) | 4 | 1 | 2 | 7
Dizziness (Nervous system disorders) | 46 | 24 | 3 | 73
Dysgeusia (Nervous system disorders) | 23 | 48 | 2 | 73
Headache (Nervous system disorders) | 123 | 86 | 8 | 214
Hypoaesthesia (Nervous system disorders) | 9 | 11 | 2 | 21
Paraesthesia (Nervous system disorders) | 17 | 18 | 0 | 35
Syncope (Nervous system disorders) | 13 | 4 | 3 | 19
Insomnia (Psychiatric disorders) | 22 | 33 | 0 | 55
Cough (Respiratory, thoracic and mediastinal disorders) | 88 | 40 | 6 | 132
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 29 | 1 | 64
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 | 6 | 4 | 41
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 | 19 | 1 | 47
Actinic keratosis (Skin and subcutaneous tissue disorders) | 10 | 24 | 2 | 36
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 138 | 0 | 164
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25 | 20 | 1 | 46
Dry skin (Skin and subcutaneous tissue disorders) | 34 | 70 | 5 | 106
Eczema (Skin and subcutaneous tissue disorders) | 28 | 13 | 4 | 45
Erythema (Skin and subcutaneous tissue disorders) | 41 | 44 | 2 | 86
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 4 | 3 | 25
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 26 | 103 | 0 | 129
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 5 | 44 | 1 | 50
Night sweats (Skin and subcutaneous tissue disorders) | 24 | 8 | 2 | 33
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 | 54 | 1 | 64
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 9 | 21 | 1 | 31
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 17 | 88 | 0 | 105
Pruritus (Skin and subcutaneous tissue disorders) | 40 | 80 | 0 | 120
Rash (Skin and subcutaneous tissue disorders) | 95 | 153 | 4 | 248
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 27 | 1 | 39
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6 | 11 | 2 | 19
Skin lesion (Skin and subcutaneous tissue disorders) | 13 | 9 | 2 | 23
Skin mass (Skin and subcutaneous tissue disorders) | 5 | 4 | 2 | 11
Hypertension (Vascular disorders) | 109 | 83 | 4 | 195
Lymphoedema (Vascular disorders) | 25 | 6 | 2 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.